CLINICAL TRIAL: NCT04327271
Title: Expanding and Scaling Two-way Texting to Reduce Unnecessary Follow-Up and Improve Adverse Event Identification Among Voluntary Medical Male Circumcision (VMMC) Clients in the Republic of South Africa
Brief Title: Two-way Texting for VMMC Follow-up in Republic of South Africa
Acronym: 2wT_RSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Aurum Institute (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Caryl Feldacker, Assistant Professor, School of Public Health, Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00009703; 1R01NR019229-01 (NIH)
Record Dates: First submitted 2020-03-20; First posted 2020-03-31 (Actual); Results first posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Voluntary Medical Male Circumcision

STUDY DESIGN:
Intervention Model Description: 2wT clients will receive automated daily texts from days 1-13. If a 2wT VMMC client responds that he suspects an AE, a VMMC nurse will exchange modifiable, scripted texts with clients to determine symptoms, frequency, and severity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text-based VMMC follow-up (Experimental): Follow-up conducted via daily text not through mandatory in person visits. Men may elect to come to the clinic if concerned about any complications but have no routine, scheduled follow-up visits.
  Interventions: Behavioral: Text-based VMMC follow-up
- Routine VMMC follow-up care (No Intervention): Routine VMMC follow up care with in person visits according to national guidelines.

INTERVENTIONS:
Behavioral: Text-based VMMC follow-up — 2wT clients will receive automated daily texts from days 1-13. If a 2wT VMMC client responds that he suspects an AE, a VMMC nurse will exchange modifiable, scripted texts with clients to determine symptoms, frequency, and severity. Then, if deemed necessary, the client will be asked to return to clinic the following day or earlier. If 2wT patients do not respond to texts or return for any visit by day 14, they will be traced by SMS, phone or home visit. All study participants will be asked to come to the clinic for study-specific, Day 14 follow-up to review healing and verify adverse event reporting. At Day 21, we will implement a brief text-based survey with 2wT clients to ascertain complete healing, providing stronger inferences at study completion.
  Arms: Text-based VMMC follow-up

SUMMARY:
Voluntary medical male circumcision (alternatively abbreviated in the literature as VMMC or MC) is a critical HIV prevention intervention with global support for expansion across sub-Saharan Africa (SSA). MC is safe: routine programs in SSA report adverse event (AE) rates well under 2%. Nevertheless, global MC guidelines require one or more follow-up visits within 14 days for AE detection. Our prior research in Zimbabwe employed two-way texting (2wT) between patients and providers to focus follow-up on men with potential AEs, allowing men healing without complication to opt-out of routine post-operative visits. 2wT safely reduced client visits by 85%, suggesting that 2wT can make MC services dramatically more efficient while maintaining safety. In the Republic of South Africa (RSA), high-volume urban clinics, remote service delivery, and low AE identification threaten quality at scale. Across more than 500,000 annual MCs performed, up to 1 million multi-stage, unnecessary MC reviews are likely conducted. RSA pressure for MC expansion and severe health system constraints, combined with good cell coverage, suggest 2wT's impact would be significant for MC care quality and efficiency, especially in rural areas. A randomized control trial (RCT) will rigorously evaluate how 2wT improves AE ascertainment and follow-up efficiency in urban and rural clinics. We aim to conduct an RCT to determine how 2wT increases AE ascertainment while reducing workload in the RSA implementation context. While the overall protocol covers multiple components over a 5-year study, this registration is specific to the RCT, aim 1.

DETAILED DESCRIPTION:
The goals and procedures overview of the randomized control trial (RCT) are to:

Generate SA evidence determining how 2wT increases AE ascertainment while reducing workload via an un-blinded, prospective, non-inferiority, RCT in urban and rural contexts comparing moderate or severe AE rate on or before the Day 14 post-MC visit and average number of in-person follow- ups control and intervention arms. For the RCT, the investigators will enroll 1104 VMMC-seeking, healthy South African men ages 18 and older in the trial, respectively, with cell phones who are seeking VMMC service at up to 5 health facilities/areas (1 urban and 4 rural) for participation in the randomized controlled study of the two-way texting (2wT) intervention. Men in the RCT will be randomly assigned 1:1 to intervention or control condition.

STUDY DESIGN RCT Study overview: The investigators will test if two-way texting (2wT) reduces unnecessary follow-up visits without compromising patient safety using a randomized control trial of 1104 men randomized 1:1 in 1 large, urban VMMC clinic and 4 rural sites clustered within one implementation team.

Study Procedures:

PARTICIPANT OVERVIEW:

• 1104 men in the full study randomized in a 1:1 ratio of texting and control for 552 men in texting and 552 in control (routine care).

1. Technology optimization
2. RECRUITMENT AND INFORMED CONSENT (RCT):

   Each site will establish local recruitment and screening methods that operationalize protocol-specified requirements for eligibility determination in a manner that is tailored to and most efficient for the local study setting and target study population. In brief, information about the study will be disseminated at the selected sites. VMMC demand creation as part of routine program practice will support study recruitment. HCW recruited for participation in the study will be reached at their workplaces (the health care facilities) following communication between the study team and the site leadership. VMMC clients will be recruited in the VMMC clinic area. Recruitment will be managed by a specifically-trained study coordinator who will meet with VMMC patients to sensitize them about the opportunity to participate in a study of text-based follow-up; those meeting eligibility criteria will be individually informed by study staff about the opportunity to participate. Interested patients will be referred to the site 2WT study coordinator. This person will meet with patients in a private setting, further explain the study, confirm study eligibility, and seek informed consent. Participant enrollment may be made by teams/clinicians using the Medic Mobile phone/tablet app or the laptop-based system.
3. RANDOMIZATION PROCESS:

   The investigators will conduct randomization using a randomized block design, ensuring that each group of 20 envelopes has 10 intervention and 10 control per block, shuffling each block to ensure a near random order. The full set of 1104 will be numbered before distribution to sites. Each group assignment envelope will be selected by the coordinator and then opened by the participant and shown to the coordinator or 2WT enrollment coordinator. Security envelopes will be used to help prevent selection of assigned group. Subjects within each block are randomly assigned to treatment conditions. This design reduces variability within treatment conditions and potential confounding, allowing for more interim analysis with near equal size groups and more certain randomization within sites.
4. Standard VMMC care (Control arm): For the 552 men randomized into the control arm, the investigators follow all NDOH protocols based on World Health Organization (WHO) guidelines including routine surgical VMMC follow-up on post-surgery days 2, 7 and 21. Patients may seek care outside scheduled visits for suspicion of AEs at any healthcare facility at any time but most often return to their VMMC site. Referral cards for VMMC clients provide local numbers for patients to text, call, or request a call back for emergencies. A standardized approach is used to assess, identify, and record the severity of AEs. All VMMC care, from assessment of all AEs through complete healing, is provided free to clients. Clients who do not return to the clinic for follow-up on Day 2 or Day 7 are considered lost to follow-up (LTFU). For the purposes of this study, control arm VMMC clients will be asked to come in on Day 14 for an additional follow-up visit. Active follow-up by phone call is provided at Day 14.
5. VMMC care procedures (2wT arm): The investigators will conduct a prospective, un-blinded, randomized control trial (RCT) among VMMC clients in a 1:1 ratio of control to intervention. Study participants and clinic staff are not masked to treatment. For the 552 men randomized into the intervention arm, men in the 2wT will receive routine VMMC surgical care and counseling, including referral cards for emergencies. 2wT clients will receive automated daily texts from days 1-13. It is free to receive call and texts; it costs approximately $0.04 to send a SMS in RSA. If they respond that they suspect no adverse event, no immediate follow-up action will be taken. If a 2wT VMMC client responds affirmatively to any daily text that he suspects an AE, a VMMC nurse will exchange modifiable, scripted texts with the client to determine the symptoms, frequency, and severity. Then, if deemed necessary, the client will be asked to return to clinic the following day or earlier if an emergency is suspected. AE management will adhere to NDOH standard care. All study participants will be asked to come to the clinic for study-specific, Day 14 follow-up to review healing and verify adverse event reporting. If 2wT patients do not respond to texts or phone and do not return on Day 14, they will be traced by SMS, Phone and up to 2 visits to their home after which they will be considered LTFU. Day 14 was chosen for verification because 95% of all AEs within a similar VMMC program in Zimbabwe are reported Day 14 or earlier, suggesting that most AEs have occurred by this time point. In a previous field study of AEs, the most common AEs of bleeding and infection were found a mean of 6.7 and 9.0 days, respectively, after VMMC, further supporting the 14 day period used in this and a previous study. The Day 14 review will be conducted by routine VMMC providers according to NDOH review guidelines. Day 14 visit may take place between days 13 and 22, depending on logistics, including patient transportation or delays.

ELIGIBILITY:
Inclusion Criteria:

For VMMC clients:

1. are at least 18 years of age or over
2. Possession of own phone at enrollment
3. Willing to respond to daily text
4. Provides contact details (phone, address)
5. Undergoes surgical MC
6. Willing to follow NDoH VMMC protocols
7. No interoperative AE
8. Informed consent
9. Receives confirmed 2wT enrollment text.

Exclusion Criteria:

For VMMC clients:

1. Not meeting above requirements
2. Men without cell phones
3. Men who chose PrePex device-based VMMC
4. Inter-operative AE during VMMC
5. No informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only men will be enrolled in the study on male circumcision. Health care workers/key informants may be male or female
Enrollment: 1093 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caryl Feldacker, PhD, MPH, Principal Investigator — University of Washington; Geoffrey Setswe, DrPH, MPH, Principal Investigator — Aurum Institute
Locations (9):
- South Africa (9):
  - Mogwase, Mogwase, Bojanala
  - Bafokeng, Phokeng, Bojanala
  - Tsakane Clinic, Brakpan, Gauteng
  - Katlehong North Clinic, Katlehong, Gauteng
  - Winnie Mandela Male Health Clinic, Tembisa, Gauteng
  - Nchabeleng Community Health Centre, Apel, Limpopo
  - Philadelphia Hospital, Dennilton, Limpopo
  - Dilokong Hospital, Driekop, Limpopo
  - Matlala Hospital, Marble Hall, Limpopo

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers.

REFERENCES:
- [Background] Feldacker C, Murenje V, Barnhart S, Xaba S, Makunike-Chikwinya B, Holeman I, Tshimanga M. Reducing provider workload while preserving patient safety via a two-way texting intervention in Zimbabwe's voluntary medical male circumcision program: study protocol for an un-blinded, prospective, non-inferiority, randomized controlled trial. Trials. 2019 Jul 23;20(1):451. doi: 10.1186/s13063-019-3470-9. PMID 31337414
- [Background] Feldacker C, Murenje V, Holeman I, Xaba S, Makunike-Chikwinya B, Korir M, Gundidza PT, Holec M, Barnhart S, Tshimanga M. Reducing Provider Workload While Preserving Patient Safety: A Randomized Control Trial Using 2-Way Texting for Postoperative Follow-up in Zimbabwe's Voluntary Medical Male Circumcision Program. J Acquir Immune Defic Syndr. 2020 Jan 1;83(1):16-23. doi: 10.1097/QAI.0000000000002198. PMID 31809358
- [Background] Feldacker C, Holeman I, Murenje V, Xaba S, Korir M, Wambua B, Makunike-Chikwinya B, Holec M, Barnhart S, Tshimanga M. Usability and acceptability of a two-way texting intervention for post-operative follow-up for voluntary medical male circumcision in Zimbabwe. PLoS One. 2020 Jun 16;15(6):e0233234. doi: 10.1371/journal.pone.0233234. eCollection 2020. PMID 32544161
- [Background] Babigumira JB, Barnhart S, Mendelsohn JM, Murenje V, Tshimanga M, Mauhy C, Holeman I, Xaba S, Holec MM, Makunike-Chikwinya B, Feldacker C. Cost-effectiveness analysis of two-way texting for post-operative follow-up in Zimbabwe's voluntary medical male circumcision program. PLoS One. 2020 Sep 30;15(9):e0239915. doi: 10.1371/journal.pone.0239915. eCollection 2020. PMID 32997710
- [Derived] Setswe G, Day S, Ndebele F, Pienaar J, Ncube V, Feldacker C. Finding the balance between rigour and relevance: implementing adaptations to the implementation of a pragmatic randomised controlled trial of a two-way texting intervention for voluntary medical male circumcision in South Africa. BMJ Open. 2025 Apr 28;15(4):e091934. doi: 10.1136/bmjopen-2024-091934. PMID 40295128
- [Derived] Feldacker C, Pienaar J, Wasunna B, Ndebele F, Khumalo C, Day S, Tweya H, Oni F, Sardini M, Adhikary B, Waweru E, Wafula MB, Dixon A, Jafa K, Su Y, Sherr K, Setswe G. Expanding the Evidence on the Safety and Efficiency of 2-Way Text Messaging-Based Telehealth for Voluntary Medical Male Circumcision Follow-up Compared With In-Person Reviews: Randomized Controlled Trial in Rural and Urban South Africa. J Med Internet Res. 2023 May 9;25:e42111. doi: 10.2196/42111. PMID 37159245
- See also: Definitions of moderate and severe adverse events from "PEPFAR's Best Practices for Voluntary Medical Male Circumcision Site Operations" — https://www.malecircumcision.org/resource/pepfar%E2%80%99s-best-practices-voluntary-medical-male-circumcision-site-operations-service-guide-0

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Text-based VMMC Follow-up | Routine VMMC Follow-up Care
Started | 553 | 540
Completed | 547 | 537
Not Completed | 6 | 3
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — randomization error (data capture) | 4 | 3

BASELINE CHARACTERISTICS:
Population: Adult men volunteering for voluntary medical male circumcision (VMMC) in South Africa
Groups:
- Total: Total of all reporting groups
Arm/Group | Text-based VMMC Follow-up | Routine VMMC Follow-up Care | Total
Number analyzed (Participants) | 553 | 540 | 1093
Age, Continuous [Mean (Full Range); unit: years] | 31.7 [18 to 61] | 31.4 [18 to 71] | 31.5 [18 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 553 | 540 | 1093
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 553 | 540 | 1093
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 553 | 540 | 1093

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Percentage of Patients With an Adverse Event (AE) (Moderate or Severe) on or Before Day 14 Visit
Description: AE rates are a global indicator of VMMC quality. This is a standard WHO and US PEPFAR government indicator as indicated in the attached reference material: PEPFAR's Best Practices for Voluntary Medical Male Circumcision Site Operations. Incidence of AEs before Day 14 will be extracted from routine VMMC data for both 2wT and control. Incident AEs on Day 14 will be identified, classified, and graded for severity using routine Ministry of Health protocols and recorded on routine VMMC AE forms. The investigators will compare cumulative rates of any moderate or severe AE on or before Day 14 between groups using Fisher's exact test as the expected number of AEs is low. The rates will be calculated per arm as: (num moderate plus severe AEs)/(total num VMMC clients who attend 2, 7 or 14 Day follow-up visit). Multivariate logistic regression models (any AE versus none) will quantify the magnitude of difference, adjusting for any potential confounders
Time Frame: Any AE before, and including, up to 22 days post VMMC to allow for logistical issues delaying attendance of the Day 14 visit
Population: The denominator is restricted to men who had at least one in-person visit before day 22 which includes the window of attendance for the D14 visit. This window also includes all AEs identified in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Text-based VMMC Follow-up | Routine VMMC Follow-up Care
Number analyzed (Participants) | 477 | 494
percentage of participants | 2.3 [1.3 to 4.1] | 1.01 [0.4 to 2.3]
Statistical Analysis 1: Comparison: Text-based VMMC Follow-up vs Routine VMMC Follow-up Care; With 10% loss to follow-up (LTFU), a sample size of 1104 men provides at least 80% power to rule out a decrease in AE ascertainment of more than 0.25% based on the lower bound of the one-sided 95% CI. The one tailed alpha was set 0.05; Test type: Non-Inferiority — Non-inferiority margin of -0.25% set as lower bound of 95% CI for the maximum mean difference between the proportion of cumulative AEs between control and 2wT arms to conclude that 2wT is non-inferior. This margin was set considering the average AE rate of 0.5% from routine SSA MC programs at scale, and assuming that 2wT increases AE ascertainment to 2.0%, similar to 1.9% of Zimbabwe RCT and the widely-accepted standard 2% AE rate; Mean Difference (Final Values) = 1.2, 95% CI 1-sided [lower limit -.09]

2. Primary Outcome: Number of Non-study In-person Visits
Description: To determine follow-up visit reduction, the investigators will compare the number of in- person visits for intervention and control using a t-test.
Time Frame: Less than or equal to 42 days post-operative
Measure: Mean (Standard Deviation); unit: Number of in-person visits
Arm/Group | Text-based VMMC Follow-up | Routine VMMC Follow-up Care
Number analyzed (Participants) | 547 | 537
Number of in-person visits | 0.22 (0.65) | 1.34 (0.85)
Statistical Analysis 1: Comparison: Text-based VMMC Follow-up vs Routine VMMC Follow-up Care; The mean number of in-person clinic visit, excluding non-study visits, were compared between the two arms using a t-test. The proportion of potential AEs was calculated as number of potential AE responses divided by the total number of daily responses (no AE and potential AE). A superiority test was performed on the safety outcomes using a two-sided 95% confidence interval and p-value using Fisher's exact test; Test type: Superiority; p = 0.001, Fisher Exact; Mean Difference (Final Values) = 1.12, 95% CI 2-sided [1.03 to 1.21]

3. Secondary Outcome: Percent of Adverse Events (AE) Identified /on/ Day 14 Visit
Description: Percentage of patients with an AE (moderate or severe) identified on the Day 14 in-person visit using AE definitions from: PEPFAR's Best Practices for Voluntary Medical Male Circumcision Site Operations
Time Frame: AEs identified during Day 14 visits that occurred only in the window between post-operative days 13-22
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Text-based VMMC Follow-up | Routine VMMC Follow-up Care
Number analyzed (Participants) | 547 | 537
percentage of participants | 0.20 [0.03 to 1.2] | 0.9 [0.4 to 2.3]

4. Secondary Outcome: Number VMMC-related Severe Adverse Events Over 22 Post-operative Days
Description: The number of severe VMMC AEs over the first 22 post operative days. The definition of "severe" in this context is any wound requiring re-opening of the wound, such as adding new sutures, from here: PEPFAR's Best Practices for Voluntary Medical Male Circumcision Site Operations. These two severe AEs were bleeding, requiring additional compression and resuturing of the wound.
Time Frame: Within 22 days post operative
Measure: Number; unit: WHO-defined severe VMMC adverse events
Arm/Group | Text-based VMMC Follow-up | Routine VMMC Follow-up Care
Number analyzed (Participants) | 547 | 537
WHO-defined severe VMMC adverse events | 2 | 0

ADVERSE EVENTS:
Time Frame: 42 post-operative days
Description: Severe and moderate adverse events defined according to, US President's Emergency Plan for AIDS Relief's (PEPFAR's) guidelines on AEs in adult voluntary medical male circumcision. AEs documented in accordance with PEPFAR guidance on routine VMMC forms. Death (suicide) not related to the study: MG1011-2351 enrolled on 10 November, 2021 and randomized to texting. No suspected AEs reported by participant. 1 December 2021 report from his work colleague of suicide on the 30th of November 2021.
Groups:
- Texting: Men who received 2-way texting (intervention)
- Routine: Routine follow-up (control)
Arm/Group | Texting | Routine
All-Cause Mortality (participants affected / at risk) | 1/547 | 0/537
Serious Adverse Events (participants affected / at risk) | 0/547 | 0/537
Other Adverse Events (participants affected / at risk) | 11/547 | 5/537
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Texting (N=547) | Routine (N=537)
Bleeding (Surgical and medical procedures) | 4 (4) | 0 (0)
Infection (Surgical and medical procedures) | 4 (4) | 2 (2)
Swelling (Surgical and medical procedures) | 0 (0) | 1 (1)
Wound disruption (Surgical and medical procedures) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
Mild AEs are not reported to the Ministry of Health nor in the study. Notifiable AEs could be underreported in either group: men could seek care for AEs at another clinic, treat themselves and not report it, or otherwise heal without intervention. Men in the 2wT arm received enhanced AE identification education with illustrative photos to explain the words of the daily response, a bias that could have increased AE identification as compared to routine. Longer term outcomes are unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT04327271/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT04327271/SAP_001.pdf
  • Informed Consent Form (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT04327271/ICF_002.pdf